CLINICAL TRIAL: NCT06729606
Title: A Multicenter, Adaptive, Randomized, Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for Hospitalized Patients With Acute Respiratory Distress Syndrome Associated With COVID-19 (Trial H1: Aviptadil)
Brief Title: Aviptadil for Severely Ill Inpatients With COVID-19 (An ACTIV-3b/TESICO Treatment Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) (Network); University of Copenhagen (Other); Medical Research Council (Other Government); Kirby Institute (Other Government); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network); US Department of Veterans Affairs (U.S. Federal Agency); Prevention and Early Treatment of Acute Lung Injury (PETAL) Network (Unknown); NeuroRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 015/ACTIV-3b/H1
Record Dates: First submitted 2024-12-10; First posted 2024-12-11 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Covid19
Keywords: COVID-19; COVID 19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; SARS-CoV-2; SARS Coronavirus; ACTIV-3; ACTIV3
MeSH Terms: conditions — COVID-19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; Severe Acute Respiratory Syndrome | interventions — aviptadil; Vasoactive Intestinal Peptide; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aviptadil + SOC (Experimental)
  Interventions: Biological: Aviptadil; Drug: Corticosteroid
- Placebo + SOC (Placebo Comparator)
  Interventions: Biological: Aviptadil Placebo; Drug: Corticosteroid

INTERVENTIONS:
Biological: Aviptadil — Administered by IV infusion over 12 hours per day for 3 days. The Day 1 infusion rate is 50 pmol/kg/hr, the Day 2 infusion rate is 100 pmol/kg/hr, and the Day 3 infusion rate is 150 pmol/kg/hr.
  Other Names: Vasoactive Intestinal Peptide; VIP
  Arms: Aviptadil + SOC
Biological: Aviptadil Placebo — Commercially available 0.9% sodium chloride solution. Administered by IV infusion over 12 hours per day for 3 days.
  Arms: Placebo + SOC
Drug: Corticosteroid — In line with NIH treatment guidelines, corticosteroids such as dexamethasone, prednisone, methylprednisolone or hydrocortisone may be administered as SOC.

SUMMARY:
This study looks at the safety and effectiveness of Aviptadil in treating COVID-19 in people who have been hospitalized with the infection and who have acute respiratory failure. Participants in the study will be treated with Aviptadil plus current standard of care (SOC), or with placebo plus current SOC.

DETAILED DESCRIPTION:
This is a treatment trial of the ACTIV-3b/TESICO master protocol (NCT04843761) to evaluate the safety and efficacy of Aviptadil at improving outcomes for patients with acute respiratory failure related to COVID-19.

This protocol will be adaptive, randomized, blinded and initially placebo-controlled. Participants will receive standard of care (SOC) treatment as part of the protocol.

This protocol will be conducted in up to several hundred clinical sites. Participating sites are affiliated with networks funded by the United States National Institutes of Health (NIH) and the US Department of Veterans Affairs.

The protocol is for a Phase 3 study.

Participants will be followed for 90 days following randomization for the primary endpoint and most secondary endpoints. Selected secondary endpoints will be measured at 180 days.

This study is planned to provide 80% power to detect an odds ratio of 1.5 for improvement in recovery status at Day 90 for Aviptadil versus placebo with use of the ordinal outcome. The planned sample size is 320 participants. Sample size may be re-estimated before enrollment is complete based on an assessment of whether the pooled proportions of the outcome are still consistent with adequate power for the hypothesized difference measured by the odds ratio.

Randomization will be stratified by study site pharmacy and by receipt of invasive mechanical ventilation, or ECMO (extracorporeal membrane oxygenation) at enrollment. Other agent-specific stratification factors may be considered.

An independent Data and Safety Monitoring Board (DSMB) will review interim safety and efficacy data at least monthly. Pre-specified guidelines will be established to recommend early stopping of the trial for evidence of harm or substantial efficacy. The DSMB may recommend discontinuation of an investigational agent if the risks are judged to outweigh the benefits.

ELIGIBILITY:
Inclusion Criteria:

Refer to the master protocol (NCT04843761)

Exclusion Criteria:

Refer to the master protocol (NCT04843761)

Additional Exclusion Criteria:

* Refractory hypotension
* Severe diarrhea
* Current C. difficile infection
* Pregnancy or current breast-feeding
* End-stage liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Brown, MD, Principal Investigator — Intermountain Medical Center/University of Utah; Prof. James Neaton, Study Chair — INSIGHT Statistical and Coordinating Centre, University of Minnesota
Locations (40):
- United States (40):
  - Banner University Medical Center Tucson (Site 206-004), 1625 N. Campbell Avenue, Tucson, Arizona
  - UCSF Fresno (Site 203-005), 155 N. Fresno Street, Fresno, California
  - VA Loma Linda Healthcare System (Site 074-017), 11201 Benton Street, Loma Linda, California
  - Cedars-Sinai Medical Center (Site 208-002), 8700 Beverly Boulevard, Los Angeles, California
  - Ronald Reagan UCLA Medical Center (Site 203-002), 757 Westwood Plaza, Los Angeles, California
  - UCSF Medical Center at Mount Zion (Site 203-007), 1600 Divisadero St., San Francisco, California
  - UCSF Medical Center (Site 203-001), Moffit-Long Hospital, 505 Parnassus Ave., San Francisco, California
  - Stanford University Hospital & Clinics (Site 203-003), 300 Pasteur Dr., Stanford, California
  - University of Colorado Hospital (Site 204-001), 12605 E. 16th Avenue, Aurora, Colorado
  - Denver Health Medical Center (Site 204-004), 780 Delaware Street, Pavilion B, Denver, Colorado
  - MedStar Health Research Institute (Site 009-021), 110 Irving St., NW., Washington D.C., District of Columbia
  - Washington DC VA Medical Center (Site 009-004), 50 Irving Street, NW., Washington D.C., District of Columbia
  - Emory University (Site 301-008), Bldg. A, Suite 2236, 1365 Clifton Rd., NE., Atlanta, Georgia
  - Massachusetts General Hospital (Site 202-002), 55 Fruit Street, Boston, Massachusetts
  - Baystate Medical Center (Site 201-001), Critical Care Research, 759 Chestnut Street, Springfield, Massachusetts
  - Mount Sinai Medical Center (Site 301-012), Icahn School of Medicine at Mount Sinai, One Gustave L. Levy Place, New York, New York
  - Columbia University Irving Medical Center (Site 301-027), 177 Fort Washington Ave., New York, New York
  - Montefiore Medical Center - Moses Hospital (Site 206-001), 111 E. 210th Street, The Bronx, New York
  - Montefiore Medical Center - Weiler campus (Site 206-003), 111 E. 210th Street, The Bronx, New York
  - Duke University Hospital (Site 301-006), 2301 Erwin Road, Durham, North Carolina
  - Wake Forest Baptist Health (Site 210-001), Medical Center Blvd, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center (Site 207-003), 234 Goodman Street, ML 0740, Cincinnati, Ohio
  - Cleveland Clinic Fairview Hospital (Site 207-005), 18101 Lorain Ave., Cleveland, Ohio
  - Cleveland Clinic Foundation (Site 207-001), 9500 Euclid Ave., Cleveland, Ohio
  - The Ohio State University Wexner Medical Center (Site 207-004), 410 W. 10th Avenue, Columbus, Ohio
  - Cleveland Clinic Marymount Campus (Site 207-006), 12300 McCracken Road, Garfield Heights, Ohio
  - Cleveland Clinic Hillcrest Hospital (Site 207-007), 6780 Mayfield Road, Mayfield Heights, Ohio
  - Oregon Health & Science University (Site 208-003), 3181 SW Sam Jackson Park Rd., Portland, Oregon
  - Medical University of South Carolina (Site 210-002), 96 Jonathan Lucas St., CSB 214, Charleston, South Carolina
  - Vanderbilt University Medical Center (Site 212-001), 1211 Medical Center Drive, Nashville, Tennessee
  - Baylor, Scott and White Health (Site 301-003), Baylor University Medical Center, 3500 Gaston Ave., Dallas, Texas
  - Houston Methodist Hospital (Site 301-028), 6565 Fannin Street, Houston, Texas
  - Texas Heart Institute (Site 301-017), 6770 Bertner, MC4-266, Houston, Texas
  - University of Texas Health Science Center (Site 203-006), 7000 Fannin St., Houston, Texas
  - Intermountain Medical Center (Site 211-001), 5121 South Cottonwood Street, Murray, Utah
  - University of Utah Hospital (Site 211-002), 50 North Medical Drive, Salt Lake City, Utah
  - UVA School of Medicine (Site 210-003), University of Virginia Health System, University Hospital, 1215 Lee St., Charlottesville, Virginia
  - Harborview Medical Center (Site 208-001), 325 9th Ave., Seattle, Washington
  - Swedish Medical Center (Site 208-005), 747 Broadway, Seattle, Washington
  - West Virginia University Medicine (Site 301-023), One Medical Center Drive, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: CDC (Centers for Disease Control and Prevention): Coronavirus (COVID-19) website — http://www.cdc.gov/coronavirus/2019-nCoV/index.html
- See also: A Participant's Guide to Clinical Trials (NIAID) — http://www.niaid.nih.gov/clinical-trials/participant-guide
- See also: Find a Clinical Trial (NIAID) — http://www.niaid.nih.gov/clinical-trials/find-a-clinical-trial
- See also: Clinical Trials at NIAID — http://www.niaid.nih.gov/clinical-trials
- See also: National Institute for Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/
- See also: WHO COVID-19 treatment guidelines — http://www.who.int/emergencies/diseases/novel-coronavirus-2019/technical-guidance/patient-management

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This substudy presents analysis for Aviptadil vs Aviptadil Placebo. Per protocol, this comparison was conducted among the pooled cohort of participants who were randomized to receive Active Aviptadil or Aviptadil Placebo within randomization strata 1, 2, and 4 of the master protocol.
Groups:
- Aviptadil + SOC: Arm includes all participants who received Aviptadil, and were randomized under strata 1, 2, and 4 from the master protocol (NCT04843761).
  Aviptadil: Administered by IV infusion over 12 hours per day for 3 days. The Day 1 infusion rate is 50 pmol/kg/hr, the Day 2 infusion rate is 100 pmol/kg/hr, and the Day 3 infusion rate is 150 pmol/kg/hr.
  Corticosteroid: In line with NIH treatment guidelines, corticosteroids such as dexamethasone, prednisone, methylprednisolone or hydrocortisone may be administered as SOC.
- Placebo + SOC: Arm includes all participants who received Aviptadil Placebo, and were randomized under strata 1, 2, and 4 from the master protocol (NCT04843761).
  Aviptadil Placebo: Commercially available 0.9% sodium chloride solution. Administered by IV infusion over 12 hours per day for 3 days.
  Corticosteroid: In line with NIH treatment guidelines, corticosteroids such as dexamethasone, prednisone, methylprednisolone or hydrocortisone may be administered as SOC.
Period: Overall Study
Arm/Group | Aviptadil + SOC | Placebo + SOC
Started | 234 | 237
Completed | 231 | 230
Not Completed | 3 | 7
Not completed — Adverse Event | 0 | 2
Not completed — Death | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Population: Number of baseline participants only include those that received an infusion.
Groups:
- Aviptadil + SOC: Arm includes all participants who received Aviptadil, and were randomized under strata 1, 2, and 4 from the master protocol (NCT04843761)
  Aviptadil: Administered by IV infusion over 12 hours per day for 3 days. The Day 1 infusion rate is 50 pmol/kg/hr, the Day 2 infusion rate is 100 pmol/kg/hr, and the Day 3 infusion rate is 150 pmol/kg/hr.
  Corticosteroid: In line with NIH treatment guidelines, corticosteroids such as dexamethasone, prednisone, methylprednisolone or hydrocortisone may be administered as SOC.
- Placebo + SOC: Arm includes all participants who received Aviptadil Placebo, and were randomized under strata 1, 2, and 4 from the master protocol (NCT04843761)
  Aviptadil Placebo: Commercially available 0.9% sodium chloride solution. Administered by IV infusion over 12 hours per day for 3 days.
  Corticosteroid: In line with NIH treatment guidelines, corticosteroids such as dexamethasone, prednisone, methylprednisolone or hydrocortisone may be administered as SOC.
- Total: Total of all reporting groups
Arm/Group | Aviptadil + SOC | Placebo + SOC | Total
Number analyzed (Participants) | 231 | 230 | 461
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 156 | 161 | 317
  >=65 years | 75 | 69 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (14.7) | 56.2 (15.1) | 56.4 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 84 | 178
  Male | 137 | 146 | 283
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 58 | 120
  Not Hispanic or Latino | 169 | 172 | 341
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 2 | 5 | 7
  Race: Asian | 7 | 10 | 17
  Race: Native Hawaiian or Pacific Islander | 3 | 3 | 6
  Race: Black or African American | 40 | 33 | 73
  Race: White | 123 | 132 | 255
  Race: More than one race | 0 | 0 | 0
  Race: Other | 16 | 11 | 27
  Race: Only ethnicity (race unknown) | 40 | 36 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 6-category Primary Ordinal Outcome (Recovery) at Day 90
Description: The primary outcome was a 6-category ordinal outcome defining the participant's status at Day 90: (1) at home (defined as the type of residence before hospitalization) and off oxygen (recovered) for at least 77 days, (2) at home and off oxygen for 49-76 days, (3) at home and off oxygen for 1-48 days, (4) not hospitalized but either on supplemental oxygen or not at home, (5) hospitalized or in hospice care, or (6) dead.
Time Frame: Status on Day 90
Population: 6 participants in the Aviptadil+SOC arm and 5 participants in the Placebo+SOC arm did not have the day 90 status available to compute the primary endpoint. These participants were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Aviptadil + SOC | Placebo + SOC
Number analyzed (Participants) | 225 | 225
Participants
  category 1 = at home and off oxygen (recovered) for at least 77 days | 36 | 31
  category 2 = at home and off oxygen for 49-76 days | 37 | 35
  category 3 = at home and off oxygen for 1-48 days | 43 | 32
  category 4 = not hospitalized but either on supplemental oxygen or not at home | 15 | 31
  category 5 = hospitalized or in hospice care | 8 | 13
  category 6 = died | 86 | 83
Statistical Analysis 1: Comparison: Aviptadil + SOC vs Placebo + SOC; Test type: Superiority; p = 0.54, Proportional odds model — Proportional odds model stratified by disease severity (high flow nasal canula [HFNC]/non-invasive ventilation [NIV] or invasive mechanical ventiliation [IMV]/ECMO) at study entry to determine the odds of being in a better category at day 90; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.80 to 1.55] — Summary odds ratio for being in a better category, active/placebo (95% confidence interval); pvalue

2. Secondary Outcome: Number of Participants Who Died Through Day 90
Time Frame: Through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Aviptadil + SOC | Placebo + SOC
Number analyzed (Participants) | 231 | 230
Participants | 86 | 83
Statistical Analysis 1: Comparison: Aviptadil + SOC vs Placebo + SOC; Test type: Superiority; p = 0.78, Cox proportional hazards model; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.77 to 1.41] — Hazard ratio for active/placebo (95% confidence interval); pvalue

3. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 5
Description: Composite safety outcome of a serious adverse event, Grade 3/4 adverse event, organ failure/serious infection, or death through Day 5
Time Frame: Through Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | Aviptadil + SOC | Placebo + SOC
Number analyzed (Participants) | 231 | 230
Participants | 146 | 129
Statistical Analysis 1: Comparison: Aviptadil + SOC vs Placebo + SOC; Test type: Superiority; p = 0.10, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.94 to 2.08] — Odds ratio for active/placebo (95% confidence interval); pvalue

4. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 28
Description: Composite safety outcome of a serious adverse event, Grade 3/4 adverse event, organ failure/serious infection, or death through Day 28
Time Frame: Through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Aviptadil + SOC | Placebo + SOC
Number analyzed (Participants) | 231 | 230
Participants | 181 | 172
Statistical Analysis 1: Comparison: Aviptadil + SOC vs Placebo + SOC; Test type: Superiority; p = 0.15, Cox proportional hazards model; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.95 to 1.44] — Hazard ratio for active/placebo (95% confidence interval); pvalue

5. Secondary Outcome: Number of Participants Who Died Through Day 180
Time Frame: Through Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Aviptadil + SOC | Placebo + SOC
Number analyzed (Participants) | 231 | 230
Participants | 90 | 86
Statistical Analysis 1: Comparison: Aviptadil + SOC vs Placebo + SOC; Test type: Superiority; p = 0.71, Cox proportional hazards model; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.79 to 1.42] — Hazard ratio for active/placebo (95% confidence interval); pvalue

ADVERSE EVENTS:
Time Frame: All-cause mortality collected through Day 180 Serious adverse events collected through Day 90 Other adverse events (not serious): Combined reporting of infusion reactions on Study days 0, 1, and 2 AND any other Adverse Events through Study Day 28.
Description: Adverse events were collected irrespective of mono or dual therapy assignment
Arm/Group | Aviptadil + SOC | Placebo + SOC
All-Cause Mortality (participants affected / at risk) | 90/231 | 86/230
Serious Adverse Events (participants affected / at risk) | 25/231 | 23/230
Other Adverse Events (participants affected / at risk) | 200/231 | 176/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aviptadil + SOC (N=231) | Placebo + SOC (N=230)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 5 (5) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Barotrauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Computerised tomogram thorax abnormal (Investigations) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aviptadil + SOC (N=231) | Placebo + SOC (N=230)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 4 (4)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0)
Acute right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 12 (13)
Bradycardia (Cardiac disorders) | 18 (21) | 22 (33)
Cardiac arrest (Cardiac disorders) | 4 (5) | 3 (3)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 2 (2)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 2 (2) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Tachycardia (Cardiac disorders) | 25 (27) | 15 (21)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye oedema (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 13 (14) | 5 (5)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (5) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8) | 7 (8)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 6 (6)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (6) | 0 (0)
Flushing (General disorders) | 34 (48) | 14 (20)
Hyperhidrosis (General disorders) | 4 (4) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 33 (49) | 31 (45)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Multisystem inflammatory syndrome (Immune system disorders) | 2 (2) | 1 (1)
Multisystem inflammatory syndrome in adults (Immune system disorders) | 0 (0) | 1 (1)
Urticaria (Immune system disorders) | 0 (0) | 2 (3)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (3) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Haemophilus bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8) | 7 (7)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 6 (6) | 4 (4)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia pseudomonal (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia staphylococcal (Infections and infestations) | 5 (5) | 7 (7)
Respiratory tract infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 5 (5)
Septic shock (Infections and infestations) | 12 (12) | 14 (16)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 4 (4)
Staphylococcal infection (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 2 (3)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Viral sepsis (Infections and infestations) | 1 (1) | 0 (0)
Barotrauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 3 (5) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (8) | 3 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (8) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Areflexia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Encephalopathy (Nervous system disorders) | 5 (5) | 4 (5)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 14 (16) | 7 (11)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 4 (4) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 4 (5) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 3 (3)
Delirium (Psychiatric disorders) | 3 (3) | 2 (2)
Intensive care unit delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 16 (19) | 22 (28)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 6 (6)
Renal impairment (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal tubular dysfunction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 14 (20) | 11 (16)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 14 (14)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (8) | 2 (3)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Endotracheal intubation (Surgical and medical procedures) | 1 (1) | 0 (0)
Haemofiltration (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal replacement therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 10 (10) | 16 (18)
Distributive shock (Vascular disorders) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 42 (61) | 38 (56)
Hypotension (Vascular disorders) | 159 (709) | 140 (687)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 6 (12)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (7):
  • Study Protocol: Aviptadil (H1) (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT06729606/Prot_007.pdf
  • Study Protocol: Remdesivir (H2) (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT06729606/Prot_011.pdf
  • Study Protocol: Master (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT06729606/Prot_012.pdf
  • Study Protocol: Overview of Study Documents (2025-08-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT06729606/Prot_013.pdf
  • Statistical Analysis Plan: Addendum (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT06729606/SAP_014.pdf
  • Statistical Analysis Plan: Main (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT06729606/SAP_015.pdf
  • Informed Consent Form (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT06729606/ICF_016.pdf